CLINICAL TRIAL: NCT00946816
Title: The Effects of Dietary Intervention on Gastrointestinal Motility, Hormonal Feedback, Visceral Sensation and Satiety in Patients With Anorexia Nervosa and Obesity
Brief Title: The Effects of Dietary Intervention on Gastrointestinal Function in Patients With Anorexia Nervosa and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Schweizerischer Nationalfonds (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNF 320030_1253331
Record Dates: First submitted 2009-07-20; First posted 2009-07-27 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Anorexia Nervosa; Obesity; Healthy Participants
MeSH Terms: conditions — Anorexia Nervosa; Obesity

ARMS (3):
- Anorexia Nervosa (Active Comparator)
  Interventions: Behavioral: Nutritional Intervention
- Obesity (Active Comparator)
  Interventions: Behavioral: Nutritional Intervention
- Healthy volunteers (Active Comparator)
  Interventions: Behavioral: Nutritional Intervention

INTERVENTIONS:
Behavioral: Nutritional Intervention — Nutritional Intervention

SUMMARY:
Diseases characterized by abnormal low and high body weight are common in the community and are associated with significant morbidity, mortality and health care related costs.

Genetic, dietary, social and psychologic factors all play an important part in these conditions; however the central role of gastrointestinal (GI) function and the control of nutrient delivery to the small bowel has not been well described in health or disease.

We propose that the GI response to feeding varies inversely with body weight. This hypothesis predicts that as body weight increases, the response to a given meal decreases in terms of motility, neurohormonal feedback, sensation and satiety. This provides an attractive explanation for why thin individuals stop eating after a small amount of food (i.e. limited gastric relaxation, rapid gastric emptying, powerful nutrient feedback with early satiety)and, conversely, why obese patients continue to eat even after nutritional requirements have been met (i.e. large gastric relaxation, slow gastric emptying, weak nutrient feedback with delayed satiety).

This project will apply MRI and Breath Tests to assess GI motility, hormonal feedback, visceral sensation and satiety in patients with pathologically low (anorexia nervosa) and high (morbid obesity) body weight and in healthy, normal weight controls.

Participants will include: Group A: normal weight, healthy volunteers (n=24: BMI: 18.5-24.9 kg/m2) Group B: patients with anorexia nervosa (DSMIV criteria and BMI: <16 kg/m2) B1: anorexia restricting type (n=12-20 over 2 years) and B2: anorexia bulimia type (n=20 over 2 years) Group C: patients with morbid obesity (BMI: 30-40 kg/m2) C1: obese (n=20 over 2 years) and C2: obese with DM type II (n=20 over 2 years).

Two studies will be performed

1. Cross-sectional study: The effects of a test meal on GI motility, hormonal feedback, visceral sensation and satiety in healthy controls and in patients with anorexia and obesity
2. Longitudinal study: The effects of dietary treatment (i.e. weight change) on GI motility, hormonal feedback, visceral sensation and satiety in patients with anorexia and obesity

ELIGIBILITY:
In addition to satisfying specific DSMIV criteria for anorexia nervosa (B1, B2) or WHO criteria for obesity (C1), or obesity and diabetes mellitus type II (C2), general inclusion criteria include:

* aged at least 18 and not more than 40 years
* able to communicate well with the investigators and provide written consent
* no physical co-morbidity requiring active treatment, in particular diabetes mellitus, impairment of liver or kidney function (subjects with diabetes mellitus type II are eligible for study group C2)
* no psychiatric (DSM IV) disorders limiting the ability to comply with study requirements
* no use of medications influencing upper GI motility within one week of the study (i.e. nitrates, prokinetic drugs, macrolide antibiotics). Acid suppression and antihypertensive medication beta-blocker, calcium channel blockers are acceptable.
* no evidence of current drug or alcohol abuse
* no history of gastrointestinal disease or surgery except appendicectomy or hernia repair
* females will take a urine pregnancy test before each study, any participant with a positive pregnancy test will be excluded (females will be investigated always in the same menstrual phase)

Exclusion criteria:

• pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The GI response to a given meal in terms of: motility, neurohormonal feedback, sensation and satiety | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fried, Professor MD, Principal Investigator — University Hospital Zurich, Gastroenterology and Hepatology
Locations (1):
- University Hospital Zurich, Gastroenterology and Hepatology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Bluemel S, Menne D, Milos G, Goetze O, Fried M, Schwizer W, Fox M, Steingoetter A. Relationship of body weight with gastrointestinal motor and sensory function: studies in anorexia nervosa and obesity. BMC Gastroenterol. 2017 Jan 5;17(1):4. doi: 10.1186/s12876-016-0560-y. PMID 28056812